CLINICAL TRIAL: NCT00574340
Title: SCCOR in Hemostatic and Thrombotic Diseases Project 5 - Metabolic Causes of Thrombosis in Type 2 Diabetes
Brief Title: Metabolic Causes of Thrombosis in Type 2 Diabetes - Question 4
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00044875-SCCOR-Q4; RFAHL04016
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Endothelial Function; Fibrinolytic Balance; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control study then antecedent hypoglycemia study group (Active Comparator): Day 1 euglycemia, day 2 hypoglycemia Hyperinsulinemic Hypoglycemic Clamp: hyperinsulinemic glucose clamp separated by 8 weeks then participants proceeded to antecedent hypoglycemia study Day 1 hypoglycemia, Day 2 hypoglycemia
  Interventions: Other: Hyperinsulinemic Hypoglycemic Clamp
- Antecedent Hypoglycemic clamp study (Active Comparator): Day 1 hypoglycemia, day 2 hypoglycemia Hyperinsulinemic Hypoglycemic Clamp: hyperinsulinemic glucose clamp separated by 8 weeks then participants proceeded to control study Day 1 euglycemia, Day 2 hypoglycemia
  Interventions: Other: Hyperinsulinemic Hypoglycemic Clamp

INTERVENTIONS:
Other: Hyperinsulinemic Hypoglycemic Clamp — all participants received (2) hyperinsulinemic glucose clamp studies separated by 8 weeks

SUMMARY:
Hypoglycemia (low blood glucose level) occurs frequently in intensively treated patients with diabetes. Although hypoglycemia was thought to occur almost exclusively in T1DM, with the advent of improved metabolic control in T2DM, the incidence of hypoglycemia is rising in these patients. Therefore in this application, we will test the novel hypothesis that prior hypoglycemia will result in (cardiovascular complications) during subsequent hypoglycemia.

DETAILED DESCRIPTION:
This study will test the hypothesis that 1) hypoglycemia causes a prothrombotic state and defective endothelial function and 2) episodes of repeated hypoglycemia will result in greater impairments of endothelial function and an increased prothrombotic tendency. Preliminary data in healthy men demonstrates that hypoglycemia can dramatically increase PAI-1 levels and the PAI-1 to tPA ratio, thereby creating a prothrombotic state. Whether this also occurs in type 2 DM patients is unknown. Furthermore, the effects of hypoglycemia on endothelial function in T2DM are also unknown.

ELIGIBILITY:
Inclusion Criteria

* 14 (7 female/ 7 male) Type 2 diabetic patients age 18-60 yrs
* 14 (7 female/ 7 male) Non-diabetic controls age and weight matched
* Body mass index >20 kg/m2
* Normal results of routine blood test to screen for hepatic, renal, and hematological abnormalities
* Female volunteers of childbearing potential: negative HCG pregnancy test
* Volunteers over 40 years old: normal baseline cardiac stress test
* For those with type 2 diabetes: HBA1C >5.5%
* For those with type 2 diabetes: diabetes < 20 years
* For those with type 2 diabetes: C-peptide >0.2 nmol (1.1-4.4 ng/ml). If c-peptide is abnormal or there is a clinical suspicion of type 1 diabetes, MODY, or LADA, Anti-Islet cell (negative) and Glutamic Acid Decarboxylase (GAD) antibody negative (0.0-1.5 U/ml) will be performed

Exclusion Criteria

* Uncontrolled hypertension
* History of cerebrovascular incidents
* Pregnancy
* Subjects unable to give voluntary informed consent
* Subjects with a recent medical illness
* Subjects on anticoagulant drugs, anemic, or with known bleeding diseases
* Tobacco Use

Physical Exam Exclusion Criteria

* Blood Pressure greater than 150/95
* Clinically significant Cardiac Abnormalities (e.g. Heart Failure, Arrhythmias, ischemic tachycardia, S-T segment deviations, ect.) from history or from cardiac stress testing
* Pneumonia
* Hepatic Failure/Jaundice
* Renal Failure
* Acute Cerebrovascular/ Neurological deficit
* Fever greater than 38.0 C

Screening blood tests exclusions according to protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Result] Joy NG, Tate DB, Younk LM, Davis SN. Effects of Acute and Antecedent Hypoglycemia on Endothelial Function and Markers of Atherothrombotic Balance in Healthy Humans. Diabetes. 2015 Jul;64(7):2571-80. doi: 10.2337/db14-1729. Epub 2015 Feb 18. PMID 25695946
- [Derived] Gogitidze Joy N, Hedrington MS, Briscoe VJ, Tate DB, Ertl AC, Davis SN. Effects of acute hypoglycemia on inflammatory and pro-atherothrombotic biomarkers in individuals with type 1 diabetes and healthy individuals. Diabetes Care. 2010 Jul;33(7):1529-35. doi: 10.2337/dc09-0354. PMID 20587723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited to participate in a cross-over design coming in for a 2 day study with an 8 week wash out period and then returning for another 2 day study. Individuals were randomized in the order of completing the control group (day 1 euglycemia, day 2 hypoglycemia) or antecedent hypo group (day 1 hypoglycemia, day 2 hypoglycemia).
Pre-assignment Details: All participants completed both studies (either the control study (day 1 euglycemia, day 2 hypoglycemia) or the antecedent hypoglycemia study (day 1 hypoglycemia, day 2 hypoglycemia) in a random order with each study separated by an 8 week wash out period.
Groups:
- Antecedent Hypoglycemia Group Then Control Study: Day 1 hypoglycemia, Day 2 hypoglycemia Hyperinsulinemic Hypoglycemic Clamp: hyperinsulinemic glucose clamp separated by 8 weeks then participants proceeded to control study Day 1 euglycemia, day 2 hypoglycemia
Period: Study 1 (2 Days)
Arm/Group | Control Study Then Antecedent Hypoglycemia Study Group | Antecedent Hypoglycemia Group Then Control Study
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Study 2 (2 Days)
Arm/Group | Control Study Then Antecedent Hypoglycemia Study Group | Antecedent Hypoglycemia Group Then Control Study
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Changes in Endothelial Function as Measured by Flow Mediated Dilation by 2D Doppler Ultrasound on Day 2
Description: A measure of the baseline arterial dilation on day 2 is compared to the post intervention measure of dilation of the brachial artery on Day 2.
Time Frame: baseline on day 2 and ~6 hours later at end of glucose clamp period
Population: Flow mediated dilation of the brachial artery
Measure: Mean (Standard Error); unit: percentage of change
Groups:
- Control Group: Day 1 euglycemia, day 2 hypoglycemia
  Hyperinsulinemic Hypoglycemic Clamp: hyperinsulinemic glucose clamp separated by 8 weeks
- Antecedent Hypoglycemia Group: Day 1 hypoglycemia, day 2 hypoglycemia
  Hyperinsulinemic Hypoglycemic Clamp: hyperinsulinemic glucose clamp separated by 8 weeks
Arm/Group | Control Group | Antecedent Hypoglycemia Group
Number analyzed (Participants) | 16 | 16
percentage of change | 2 (1) | 7 (1)

ADVERSE EVENTS:
Time Frame: 1 year or until study participation was completed.
Groups:
- Control Group- All Participants: Day 1 euglycemia, day 2 hypoglycemia= one study
  Hyperinsulinemic Euglycemic Clamp study: each two day study (arm) separated by 8 weeks
- Antecedent Hypoglycemia Group-all Participants: Day 1 hypoglycemia, day 2 hypoglycemia= one study
  Hyperinsulinemic Hypoglycemic Clamp study: each two day study (arm) separated by 8 weeks
Arm/Group | Control Group- All Participants | Antecedent Hypoglycemia Group-all Participants
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No